CLINICAL TRIAL: NCT02612116
Title: The Impact of Administration Strategy of Ticagrelor on Its Pharmacokinetics and Pharmacodynamics in Patients With Unstable Angina Pectoris - a Randomized, Single-center, Open-label Pilot Study
Brief Title: Comparison of Administration Strategies of Ticagrelor in Patients With Unstable Angina Pectoris, a Pharmacokinetic / Pharmacodynamic Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Collegium Medicum w Bydgoszczy (Other)
Responsible Party: Principal Investigator, Jacek Kubica, Prof. Jacek Kubica, MD, PhD, Collegium Medicum w Bydgoszczy
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CMUMK202D
Record Dates: First submitted 2015-11-19; First posted 2015-11-23 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Unstable Angina Pectoris
MeSH Terms: conditions — Angina, Unstable | interventions — Ticagrelor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- pulverized ticagrelor sublingually (Active Comparator): Pulverized ticagrelor 180 mg (Brilique) administered sublingually
  Interventions: Drug: Pulverized ticagrelor sublingually
- pulverized ticagrelor orally (Active Comparator): Pulverized ticagrelor 180 mg (Brilique) administered orally
  Interventions: Drug: Pulverized ticagrelor orally
- Integral ticagrelor orally (Active Comparator): Ticagrelor 180 mg (Brilique) administered orally in integral tablets
  Interventions: Drug: Integral ticagrelor

INTERVENTIONS:
Drug: Pulverized ticagrelor sublingually — Pulverized ticagrelor (180 mg) administered sublingually
  Other Names: Brilique
  Arms: pulverized ticagrelor sublingually
Drug: Pulverized ticagrelor orally — Pulverized ticagrelor (180 mg) administered orally
  Other Names: Brilique
  Arms: pulverized ticagrelor orally
Drug: Integral ticagrelor — Integral ticagrelor (180 mg) administered orally
  Other Names: Brilique
  Arms: Integral ticagrelor orally

SUMMARY:
The purpose of this study is to evaluate the differences in pharmacokinetics and pharmacodynamics of ticagrelor and its active metabolite depending on the strategy of the drug administration in patients with unstable angina pectoris.

DETAILED DESCRIPTION:
On the basis of the current guidelines ticagrelor is a recommended antiplatelet agent in acute coronary syndromes, including unstable angina pectoris.

According to the results of the MOJITO study, performed in patients with ST-elevation myocardial infarction, the effect of ticagrelor, measured as platelet inhibition, may be achieved sooner when crushed tablets are administered. Thus, there may be significant differences in pharmacokinetics and pharmacodynamics of ticagrelor if pulverized drug is given orally or sublingually when compared with currently used oral administration of integral tablets.

The study is designed as an open-label, single-center, randomized trial of different strategies of administration of ticagrelor in patients with unstable angina pectoris. After enrollment, the participants will be randomized into three arms, each receiving ticagrelor. The drug will be given in: (1) pulverized tablets administered sublingually, (2) pulverized tablets administered orally or in (3) integral tablets orally. The time required for ticagrelor and its active metabolite AR-C124900XX to reach their maximum serum concentration will be measured as the primary outcome of the study. Moreover, further evaluation of other parameters including maximum plasma concentration and area under the plasma concentration of ticagrelor and its active metabolite will be assessed as secondary outcomes. The platelet reactivity will be measured with the Multiplate Analyzer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent prior to any study specific procedures
* Diagnosis of unstable angina
* Male or non-pregnant female, aged 18-80 years old
* Provision of informed consent for angiography and percutaneous coronary intervention (PCI)
* GRACE score <140 pts

Exclusion Criteria:

* treatment with ticlopidine, clopidogrel, prasugrel or ticagrelor within 14 days before the study enrollment
* hypersensitivity to ticagrelor
* current treatment with oral anticoagulant or chronic therapy with low-molecular-weight heparin
* active bleeding
* history of intracranial hemorrhage
* recent gastrointestinal bleeding (within 30 days)
* history of coagulation disorders
* platelet count less than <100 x10^3/mcl
* hemoglobin concentration less than 10.0 g/dl
* history of moderate or severe hepatic impairment
* history of major surgery or severe trauma (within 3 months)
* patients considered by the investigator to be at risk of bradycardic events
* second or third degree atrioventricular block during screening for eligibility
* history of asthma or severe chronic obstructive pulmonary disease
* patient requiring dialysis
* manifest infection or inflammatory state
* Killip class III or IV during screening for eligibility
* respiratory failure
* history of severe chronic heart failure (NYHA class III or IV)
* concomitant therapy with strong CYP3A inhibitors (ketoconazole, itraconazole, voriconazole, telithromycin, clarithromycin, nefazadone, ritonavir, saquinavir, nelfinavir, indinavir, atazanavir) or strong CYP3A inducers (rifampicin, phenytoin, carbamazepine, dexamethasone, phenobarbital) within 14 days and during study treatment
* body weight below 50 kg

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2015-09; Primary Completion 2016-08 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Time to maximum concentration (tmax) for ticagrelor and AR-C124900XX | 6 hours

SECONDARY OUTCOMES:
Maximum ticagrelor and AR-C124900XX concentration | 6 hours
Area under the plasma concentration-time curve for ticagrelor (AUC 0-6h) | prior to the initial dose and 15 min, 30 min, 45 min, 1, 2, 3, 4, 6 hours post dose
Area under the plasma concentration-time curve for AR-C124900XX (AUC 0-6h) | prior to the initial dose and 15 min, 30 min, 45 min, 1, 2, 3, 4, 6 hours post dose
Platelet reactivity assessed by Multiple Electrode Aggregometry | prior to the initial dose and 30min, 1, 2, 3, 4, 6 hours post dose

CONTACTS AND LOCATIONS:
Overall Officials: Jacek Kubica, MD., PhD., Principal Investigator — Cardiology Department, Dr. A. Jurasz University Hospital
Locations (1):
- Cardiology Department, Dr. A. Jurasz University Hospital, Bydgoszcz, Kuyavian-Pomeranian Voivodeship, Poland